CLINICAL TRIAL: NCT00453895
Title: Sunitinib in Refractory Adrenocortical-Carcinoma Patients Progressing After Cytotoxic Chemotherapy
Brief Title: Sunitinib in Refractory Adrenocortical Carcinoma
Acronym: SIRAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Martin Fassnacht, Professor for Medicine and Endocrinology, University of Wuerzburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIRAC-1
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenal cancer refractory to cytotoxic therapy; Sunitinib; Multitargeted tyrosine-kinase inhibitor
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib (Experimental): Sunitinib will be administered 50 mg per day for 4 weeks followed by 2 weeks off.
  treatment will continue until progressive disease or unacceptable toxicity
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50mg Sunitinib

SUMMARY:
Although a first randomized trial in patients with advanced ACC leading to the establishment of a first line cytotoxic chemotherapy is ongoing (FIRM-ACT), the failure rate even of this FIRM-ACT study is most likely clearly above 50%. Therefore, the majority of participating patients urgently need a new treatment option. However, up to date there is no evidence for a single regimen that might be promising in these treatment-refractory patients with ACC.

Sunitinib is an oral multitargeted tyrosine kinase inhibitor with anti-tumor and antiangiogenic activities, which is successfully tested in the treatment of patients with metastatic renal cell carcinoma, gastrointestinal stromal and neuroendocrine tumors after failure of standard cytotoxic chemotherapy.

The primary objective of this trial is to estimate the response (defined as progression-free survival of ≥ 12 weeks) rate associated with Sunitinib treatment in patients advanced ACC progressing after cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ACC
* Locally advanced or metastatic disease not amenable to radical surgery resection
* Radiologically monitorable disease
* Progressing disease after one to three cytotoxic chemotherapy regimes including a platin-based protocol
* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Age ≥ 18 years
* Adequate bone marrow reserve (neutrophils ≥ 1500/mm³ and platelets ≥100.000/mm³) and haemoglobin ≥ 9 g/dl
* Negative pregnancy test and effective contraception in pre-menopausal female and male patients
* Patient´s written informed consent
* Ability to comply with the protocol procedures
* If patients have been participated in another clinical trial evaluating treatment options for ACC (e.g. FIRM-ACT), the patient can only be included in the SIRAC trial, if:

  * the patient has discontinued study treatment of the previous trial according to the protocol
  * or the study chair of the previous trial gives written approval for inclusion of this individual patient in the SIRAC trial.

Exclusion Criteria:

* History of prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years.
* Severe renal (serum creatinine > 2.5 x ULN) or hepatic insufficiency (ALT / AST > 2.5 x ULN or ALT/AST >5 x ULN if liver function abnormalities are due to the underlying malignancy and/or total serum bilirubin > 2.0 x ULN) and/or serum albumin < 3g/dl
* Any of the following within the 8 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, or other severe thromboembolic event.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade 2, acute atrial fibrillation of any grade, or prolongation of the QTc interval to >470 msec for females
* Left ventricular ejection fraction (LVEF) <45% as measured by echocardiogram
* NCI CTCAE Grade 3 hemorrhage within 4 weeks of starting study treatment
* Hypertension that cannot be controlled by medications (>160/100 mmHg despite optimal medical therapy)
* Pregnancy or breast feeding
* Previous treatment with Sunitinib or any other VEGF- or PDGF-pathway directed agent.
* Current treatment with strong CYP3A4 inhibitors or -inducers
* Current treatment with another investigational drug
* Current treatment with another anti-cancer drug
* Patients with ileus within the last 28 days
* Major surgery, radiation therapy, or systemic therapy within 3 weeks of first study treatment. At least 7 days should elapse from the time of minor surgical procedure including placement of an access device or fine needle aspiration before start of study treatment
* Serious wounds that have not completely healed, active ulcer(s), or significant bone fracture(s).
* Prior radiation therapy to >25% of the bone marrow.
* Cachectic patients with a body mass index < 18 kg/m2
* Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-07; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fassnacht, MD, Principal Investigator — University of Wuerzburg
Locations (2):
- Germany (2):
  - Charite Berlin, Berlin
  - Dept. of Medicine I, University of Wuerzburg, Würzburg

REFERENCES:
- [Result] Kroiss M, Quinkler M, Johanssen S, van Erp NP, Lankheet N, Pollinger A, Laubner K, Strasburger CJ, Hahner S, Muller HH, Allolio B, Fassnacht M. Sunitinib in refractory adrenocortical carcinoma: a phase II, single-arm, open-label trial. J Clin Endocrinol Metab. 2012 Oct;97(10):3495-503. doi: 10.1210/jc.2012-1419. Epub 2012 Jul 26. PMID 22837187

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was included in the study on July 17, 2007, the last patient enrolled on September 18, 2009. The last patient stopped the study drug on November 20, 2009.
Groups:
- Sunitinib: Sunitinib will be administered 50 mg per day for 4 weeks followed by 2 weeks off.
  treatment will continue until progressive disease or unacceptable toxicity
  Sunitinib :
Period: Overall Study
Arm/Group | Sunitinib
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 17
Region of Enrollment [Number; unit: participants]
  Germany | 39

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Clinical Benefit Due to Treatment With Sunitinib
Description: Clinical benefit was defined as stable disease or better for at least 12 weeks
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 35
Participants | 5

2. Secondary Outcome: Assessment of Objective Response Rates
Description: Objective Response Rate defined by RECIST 1.0
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 35
Participants | 0

3. Secondary Outcome: Assessment of Progression-free Survival
Description: Progression-free survival is defined as time of start of study until documentation of Progress. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: up to 400 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sunitinib
Number analyzed (Participants) | 35
days | 83 [80 to 85]

4. Secondary Outcome: Assessment of Overall Survival
Description: Overall Survival was defined as time from start of treatment until death or last follow-up.
Time Frame: up to 36 months
Measure: Median (95% Confidence Interval); unit: monhts
Arm/Group | Sunitinib
Number analyzed (Participants) | 35
monhts | 5.4 [3.2 to 7.6]

5. Secondary Outcome: Assessment of Toxicity
Description: Adverse events were rated using the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 (see http://ctep.cancer.gov/reporting/ctc.html).
Time Frame: up to 400 days
Measure: Median (Full Range); unit: number of adverse events/patient
Arm/Group | Sunitinib
Number analyzed (Participants) | 39
number of adverse events/patient | 4 [0 to 10]

ADVERSE EVENTS:
Time Frame: up to 1 year
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 10/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=39)
myocard infarcton (Cardiac disorders) | 1 (1)
hypogylcimia (Endocrine disorders) | 1 (1)
Dizziness/drowsiness (Nervous system disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
liver failure (General disorders) | 1 (1)
adrenal insufficiency (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=39)
Polyneuropathy (Nervous system disorders) | 10 (11)
Pain (General disorders) | 10 (15)
Diarrhea (Gastrointestinal disorders) | 9 (9)
rash or discolored nails (Skin and subcutaneous tissue disorders) | 9 (9)
fatigue (General disorders) | 3 (3)
mucositis (Skin and subcutaneous tissue disorders) | 4 (4)
Anemia, Thrombopenia, Leukopenia (Blood and lymphatic system disorders) | 4 (4)
hemorrhage (Blood and lymphatic system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
A limitation arises from the fact that imaging prior study entry was not standardized. Therefore we cannot provide data regarding the dynamics of tumor growth before initiation of sunitinib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes